CLINICAL TRIAL: NCT05633901
Title: Evaluation of Preoperative Counseling Video on Anxiety in Patients Undergoing Vaginal Prolapse Surgery
Brief Title: Impact of Preop Video on Patient Anxiety
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22-094
Record Dates: First submitted 2022-11-07; First posted 2022-12-01 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Prolapse, Vaginal; Prolapse, Uterine; Prolapse; Female
Keywords: Anxiety; Video; Prolapse; Urogynecology
MeSH Terms: conditions — Uterine Prolapse; Prolapse; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Placebo Comparator): Standard verbal counseling provided to patients by clinic nurse about post-operative expectations
  Interventions: Other: Standard Counseling
- Educational Video (Active Comparator): An educational video to aid standard counseling packet on post-operative expectations
  Interventions: Other: Educational Video

INTERVENTIONS:
Other: Educational Video — Patients will be given the link to the educational video and able to view it as many times as they want
  Arms: Educational Video
Other: Standard Counseling — Current standard of care verbal counseling from a clinic nurse
  Arms: Standard of Care

SUMMARY:
To determine whether a pre-operative educational video has an impact on the anxiety of patients undergoing vaginal prolapse surgery

ELIGIBILITY:
Inclusion Criteria:

* Prolapse surgery may include: apical repair with uterosacral ligament suspension, or sacrospinous/iliococcygeal ligament fixation, or sacrocolpopexy.
* They may also have a concomitant total vaginal hysterectomy with or without bilateral salpingectomy/oophorectomy, other compartment repairs for prolapse, or a suburethral sling for incontinence.
* Surgery by one of the fellowship trained Urogynecologists at TriHealth
* Age >= 18
* English speaking
* Able to comprehend and answer the survey completely.

Exclusion Criteria:

* Concomitant procedure with another surgeon
* Resides in a nursing home
* Non-English speaking
* Patients with mental disability, Alzheimer's disease, dementia that would preclude complete answering of the survey or inability to answer the questions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Pre-operative anxiety level in each group, as measured with the Surgical Anxiety Questionnaire. | Immediately Pre-op
  Surgical Anxiety Questionnaire is a validated, 17 question survey with scores ranging from 0 (least anxious) to 68 (most anxious)

SECONDARY OUTCOMES:
To assess a difference in anxiety levels, based on Surgical Anxiety Questionnaire score, in patients currently taking medication for anxiety | Immediately Pre-op
  Surgical Anxiety Questionnaire is a validated, 17 question survey with scores ranging from 0 (least anxious) to 68 (most anxious)
To assess a difference in anxiety levels, based on Surgical Anxiety Questionnaire score, in patients that did or did not watch the video at home | Immediately Pre-op
  Surgical Anxiety Questionnaire is a validated, 17 question survey with scores ranging from 0 (least anxious) to 68 (most anxious)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cincinnati Urogynecology Associates, Cincinnati, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No